CLINICAL TRIAL: NCT01418404
Title: The Application of Thermal Stimulation on Functional Recovery of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: E-DA Hospital (Other); Kaohsiung Municipal Hsiaokang Hospital (Other Government)
Responsible Party: Principal Investigator, Jau-Hong Lin, Professor, Professor in Department of Physical Therapy, Kaohsiung Medical University, Taiwan, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NHRI-EX99-9907PI
Record Dates: First submitted 2011-06-26; First posted 2011-08-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: Stroke; Effects of TS in U/E motor recovery; Brain mapping; Kinematics analysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Noxious TS in study A (Experimental): Noxious TS in study A
  Interventions: Other: Noxious TS
- Innocuous TS (Active Comparator): Innocuous TS in study A
  Interventions: Other: Innocuous TS
- High Frequency of Noxious TS (Experimental): High Frequency of Noxious TS in study B
  Interventions: Other: High Frequency of Noxious TS
- Low Frequency of Noxious TS (Active Comparator): Low Frequency of Noxious TS in study B
  Interventions: Other: Low Frequency of Noxious TS
- High Intensity of Noxious TS (Experimental): High Intensity of Noxious TS in study C
  Interventions: Other: High Intensity of Noxious TS
- Low Intensity of Noxious TS (Active Comparator): Low Intensity of Noxious TS in study C
  Interventions: Other: Low Intensity of Noxious TS

INTERVENTIONS:
Other: Noxious TS — hot, cold alternately, noxious TS in study A
  Arms: Noxious TS in study A
Other: Innocuous TS — warm, cool alternately, Innocuious TS in study A
  Arms: Innocuous TS
Other: High Frequency of Noxious TS — High Frequency of Noxious TS in study B
  Arms: High Frequency of Noxious TS
Other: Low Frequency of Noxious TS — Low Frequency of Noxious TS in study B
  Arms: Low Frequency of Noxious TS
Other: High Intensity of Noxious TS — High Intensity of Noxious TS in study C
  Arms: High Intensity of Noxious TS
Other: Low Intensity of Noxious TS — Low Intensity of Noxious TS in study C
  Arms: Low Intensity of Noxious TS

SUMMARY:
In literature review, thermal stimulation (TS) intervention is effective in facilitating upper extremity functional recovery in stroke patients. In addition, several functional MRI studies have indicated that thermal stimuli promoted activation in the premotor and motor cortices of healthy participants. These imply the possibility of TS in cortical reorganization. However, there were no studies exploring the relationship of the TS intervention and cortical reorganization. By the functional recovery of stroke patients, findings of brain image and brain mapping, it could enhance the understanding the TS influences on brain reorganization. Regarding with clinical application of the TS intervention for improving functional performance of upper extremity in participants with stroke, the best parameters of TS intervention in clinical practice have not been decided. Therefore, this five-year study recruited three groups of stroke patients (acute, sub-acute, chronic) undergoing TS intervention with different parameters. Functional scales, kinematic data, brain image were taken in several timelines as outcome measures.

DETAILED DESCRIPTION:
The thermal stimulation (TS) intervention uses the heat and cold apply alternately (~30minutes), and this kind temperature application is common in clinical neuromuscular or sports rehabilitation. Moreover, some studies have proved efficacy of the TS on stroke. However, the best parameters and application on different-stage stroke groups have not been clearly explored. Moreover, in order to discover the TS intervention influences on neuroplasticity, the brain images and the brain mapping are taken in the group A (explained in the below). In addition, the kinematic data was also collected in group A. However, the above-mentioned three examination are optional. Finally, functional recovery measurements (clinical scales) are measured in the three groups.

There are three groups (90 participants in each group) and their respective TS intervention design. In other word, three sub-studies (A, B, C) are under this project. Group A recruited 90 acute stroke (~ 30 days) and the independent variable is temperature of TS intervention. Group B is with sub-acute stroke (3-12 months), undergoing different frequency of TS intervention. Group C targets on participants with chronic stroke (> 1 y/o) and this variation in TS is intensity of TS application (30 mins vs 60 mins/each session).

ELIGIBILITY:
Inclusion Criteria:

1. first-ever ischemic stroke;
2. no severe cognitive impairments and able to follow instructions;
3. sit on a chair for more than 30 minutes independently.

Exclusion Criteria:

1. musculoskeletal or cardiac disorders that potentially interferes with experimental tests;
2. diabetic or sensory impairment that attributable to peripheral vascular disease or neuropathy;
3. speech disorder or global aphasia;
4. skin problems at the sites of stimulation;

6.contraindications of heat or ice application.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Movement performance assessment | baseline, half time-line of whole intervention period, post-intervention, 1 month follow-up, 6 month follow-up
  * Movement performance assessment by clinical motor assessment scales in upper extremity
  * executed by qualified physiotherapy
  * in study A, B, C
Brain images | immediate effects in 3 timeline
  * "intermediate effect of TS" means: pretest of the single TS, then application of this single TS, finally post-test of this TS in the session in the same day
  * immediate effects of intervention in the 1st day and 24th of intervention, six-month follow-up
  * this examination is optional
  * in study A.
  * use regular scan examination of hospital and operated by trained qualified professionals, the attending is consulted
  * This examination can be stopped at any time if participants do not want to perform or feeling unwell
Mapping of brain cortex | immediate effect in four timeline
  * "intermediate effect of TS" means: pretest of the single TS, then application of this single TS, finally post-test of this TS in the session in the same day
  * immediate effects of intervention in the 1st day and 24th of intervention, one-month follow-up, six-month follow-up
  * in study A.
  * this examination is optional
  * use equipment of brain mapping and operated under trained staff, the attending is consulted This examination can be stopped at any time if participants do not want to perform or feeling unwell
Kinematics measure of upper extremity movement | four timeline
  * 1st day and 24th of intervention, one-month follow-up, six-month follow-up (This examination is optional)
  * signal emission marks are sticked on surface skin during motion tests
  * this examination is optional
    --in study A.
  * executed by trained qualified physiotherapy

SECONDARY OUTCOMES:
Quality of life | baseline, post-intervention, 6 month follow-up
  * Quality of life by subjective questionnaires
  * executed by qualified physiotherapy --in study A, B, C.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Hong Lin, Professor, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan, Taiwan

REFERENCES:
- [Derived] Chen SC, Hsu MJ, Kuo YT, Lin RT, Lo SK, Lin JH. Immediate effects of noxious and innocuous thermal stimulation on brain activation in patients with stroke. Medicine (Baltimore). 2020 Feb;99(9):e19386. doi: 10.1097/MD.0000000000019386. PMID 32118788